CLINICAL TRIAL: NCT00647322
Title: The Impact of Reducing Overtreatment on Quality of Life in Children With Refractory Epilepsy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Child Health (Other)
Responsible Party: R&D Office, Institute of Child Health
Allocation: Non-Randomized | Model: Single Group | Masking: Single
Other Study IDs: 07NR07
Record Dates: First submitted 2008-03-26; First posted 2008-03-31 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: Intractable Epilepsy
Keywords: Intractable epilepsy, Drug Reduction, Antiepileptic medication
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- 1 (Experimental): Reduction in anti-epileptic medications
  Interventions: Other: Reduction of anti-epileptic medications
- 2 (Active Comparator): No change in medication. Unchanged treatment
  Interventions: Procedure: No drug change

INTERVENTIONS:
Other: Reduction of anti-epileptic medications — Reduction in anti-epileptic medications
  Arms: 1
Procedure: No drug change — No change in anti-epileptic treatment
  Arms: 2

SUMMARY:
The primary aim of the study is to determine the effect of reducing the number and/or dose of anti epileptic drugs on an individual's quality of life and seizure control in people with difficult to control epilepsy and who are on polytherapy.

This is a randomised trial so children will be divided into two groups, with reduction of anti epileptic drugs in the first group (withdrawal group) and no change to their medications in the second (control group). Irrespective of the group the child is assigned to (withdrawal group or control group), we will ask parents to complete several questionnaires on 2 occasions: the first time will be immediately after the child enters the study (i.e. baseline assessment), and a second and last one will be 6 months after entering the study (i.e. follow-up assessment). These questionnaires aim to "quantify" aspects related with quality of life, AED side effects, seizure severity, and behaviour.

ELIGIBILITY:
Inclusion Criteria:

* Young people aged 6-21 years with intractable epilepsy receiving antiepileptic drug polytherapy

Exclusion Criteria:

* None

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2008-09; Primary Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Effect of reduction in anti-epileptic medications on quality of life in young people with intractable epilepsy | 6 months

SECONDARY OUTCOMES:
Identify other determinants of quality of life in this group of subjects | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Neurosciences Unit, UCL Institute of Child Health, The Wolfson Centre,, London, United Kingdom